CLINICAL TRIAL: NCT02601443
Title: Prevention of Preterm Birth With a Pessary in Triplet
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: never started
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 213/15
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Pessary (Experimental): Cervical pessary is a medical device used to treat an incompetent (or insufficient) cervix (cervix starts to shorten and open too early). Early in the pregnancy a round silicone pessary is placed at the opening to the cervix to close it, and then remove late in the pregnancy when the risk of a preterm birth has passed.
  Cervical pessary has been tried as a simple, non-invasive alternative that might replace the above invasive cervical stitch operation to prevent preterm birth.
  Interventions: Device: Cervical Pessary
- Routine care (watch and wait) (No Intervention)

INTERVENTIONS:
Device: Cervical Pessary
  Arms: Cervical Pessary

SUMMARY:
The incidence of multiple gestations has increased over the past years, mostly because of increased use of assisted reproductive technologies. Triplet pregnancies are at increased risk of preterm birth (PTB), which is the primary reason for their increased morbidity and mortality compared to singletons. Multiple gestations, including triplets, account for about 3% of all pregnancies in the US but constitute at least 10% of cases of PTB, over 30% of very low birth weight infants, and nearly 20% of infant mortality.

A short cervical length (CL) on transvaginal ultrasound (TVU) has been shown to be a good predictor of PTB, including in multiple gestations. In singletons with a prior PTB and a short CL <25mm before 24weeks, cerclage is associated with significant decreases in PTB and perinatal morbidity and mortality in the meta-analysis of randomized trials (RCTs). On the contrary, the effect of cerclage in multiple gesttations has been insufficiently studied, with meta-analysis data showing a possible harm from cerclage compared to controls.

The aim of this RCT is to evaluate the efficacy of cervical pessary in prevention of PTB in unselected triplet gestations.

We planned to assess outcomes in subgroup analysis of women with short cervical length (TVU CL <30 mm)

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Triplet pregnancy (limits the participants to female gender)
* Gestational age at randomization between 20(0) and 22(6)

Exclusion Criteria:

* Singleton, twin or higher order than triplets multiple gestation
* Twin twin transfusion syndrome
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Cerclage in place (or planned placement)
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina
* Painful regular uterine contractions
* Labor
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery | Less than 34 weeks gestation

SECONDARY OUTCOMES:
Gestational age at delivery | Time of delivery
Birth weight | Time of delivery
pontaneous preterm birth rates | Less than 24, 28, 34 and 37 weeks gestation
Spontaneous rupture of membranes | Less than 34 weeks gestation
Type of delivery: rate of cesaran delivery, vaginal delivery and operative vaginal delivery | Time of delivery
Neonatal death | Between birth and 28 days of age
Composite adverse neonatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia (BPD), retinopathy, blood-culture proven sepsis and neonatal death
Admission to neonatal intensive care unit | Between birth and 28 days of age
Chorioamnionitis | Time of delivery
Significant adverse maternal effects | Time of delivery
  Includes heavy bleeding, injury (eg erosion; fistula; etc) to vagina; injury (eg erosion; fistula; etc) to bladder, cervical tear and uterine rupture
Intolerance to pessary | Prior to delivery
  Defined as request for removal secondary to discomfort and/or discharge
Preterm delivery | Less than 24, 28 and 37 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Naples, Italy